CLINICAL TRIAL: NCT05280236
Title: Comparison of Quality of Recovery Between Remimazolam and Propofol Anesthesia in Patients Undergoing Arthroscopic Meniscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2021-1803
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Adult Patients 19 or Older Scheduled for Elective Arthroscopic Meniscectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Patients receiving general anesthesia with propofol-based total intravenous anesthesia
  Interventions: Drug: Propofol TIVA
- Remimazolam (Experimental): Patients receiving general anesthesia with remimazolam-based total intravenous anesthesia
  Interventions: Drug: Remimazolam TIVA

INTERVENTIONS:
Drug: Propofol TIVA — Patients will receive propofol-based TIVA with propofol and remifentanil TCI (target controlled infusion)
  Arms: Propofol
Drug: Remimazolam TIVA — Patients will receive remimazolam-based TIVA with remimazolam infusion and remifentanil TCI
  Arms: Remimazolam

SUMMARY:
This study aims to compare quality of recovery after surgery and anesthesia between patients undergoing arthroscopic meniscectomy under general anesthesia with either propofol or remimazolam based total intravenous anesthesia. This study is a randomized trial with a 50% probability of being assigned to either group. Randomization will be done by an anesthesiologist not involved in anesthesia or postoperative outcome assessment. Patients and the investigator in charge of postoperative outcomes assessment will be blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 19 or older, ASA class I~III,
* scheduled for arthroscopic meniscectomy under general anesthesia and eligible for LMA use.

Exclusion Criteria:

* Patient refusal,
* patients unable to read consent form, active URI or uncontrolled asthma,
* pneumonia,
* history of allergies to propofol or benzodiazepines,
* decreased liver or kidney function, heart failure of ejection fraction<55%,
* pregnant or breastfeeding patients,
* history of substance abuse/addiction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery (QoR)-40 questionnaire | Postoperative 24 hours
  Quality of recovery assessed with the QoR-40 questionnaire, which is a widely-used, self-rated, self-completed questionnaire for postoperative patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No